CLINICAL TRIAL: NCT07190469
Title: A Phase 1, Open-label, Multicenter Clinical Trial Evaluating the Safety, Pharmacokinetics, Pharmacodynamics and Anti-Cancer Activity of PQ203 in Patients With Advanced Solid Tumor Malignancies
Brief Title: PQ203 in Advanced Malignant Tumors Including Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ProteinQure Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PQ203-001
Record Dates: First submitted 2025-08-19; First posted 2025-09-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Triple Negative Breast Cancer (TNBC); Advanced Solid Tumors Cancer
Keywords: Triple Negative Breast Cancer; TNBC; PQ203; advanced solid tumors; Phase 1
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PQ203 (Experimental): A Phase 1, first-in-human (FIH), multiple ascending dose study of the peptide drug-conjugate PQ203 to evaluate the safety, pharmacokinetics, tolerability and preliminary anti-cancer activity in patients with advanced cancers with solid tumors. Comprises up to 7 planned ascending dose cohorts with expansion of doses to identify recommended dose levels for testing in the Phase 1B Dose Optimization study. This is an open label study and all participants will receive PQ203.
  Interventions: Drug: PQ203

INTERVENTIONS:
Drug: PQ203 — PQ203 is a peptide drug-conjugate given once weekly by intravenous infusion intended for the treatment of advanced solid tumor cancers including triple negative breast cancer.

SUMMARY:
The primary purposes of this study are to determine the safety and tolerability of PQ203 in patients with advanced solid tumors including triple negative breast cancer (TNBC), and to determine a recommended Phase 2 dose level for future studies in TNBC.

DETAILED DESCRIPTION:
This is an open-label, first-in-human study designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of PQ203 in patients with selected advanced solid tumors. PQ203 will be administered as a once-weekly intravenous infusion.

The study consists of two parts: Phase 1A (dose escalation/expansion) and Phase 1B (dose optimization).

* Phase 1A will employ a dose-escalation design in patients with advanced solid tumors to assess the safety and tolerability of PQ203 as monotherapy and to establish a provisional Recommended Phase 2 Dose (RP2D). A dose-expansion component will further evaluate the provisional RP2D in one or more selected tumor types.
* Phase 1B will assess the provisional RP2D and further characterize safety, pharmacokinetics, and preliminary efficacy.

Endpoints:

* Primary Endpoints: Incidence of treatment-emergent adverse events (TEAEs) and determination of the RP2D.
* Secondary Endpoints: Pharmacokinetic profile of PQ203 and its payload (MMAE), and preliminary evidence of antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Histologically or cytologically documented metastatic or locally advanced solid tumor malignancies having progressed through or being otherwise ineligible to receive approved standard-of-care therapies
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Documented presence of RECIST v1.1 measurable disease
* Adequate organ function confirmed by the following laboratory values obtained within 14 days of the first dose of PQ203:

Bone Marrow Function

* Absolute neutrophil count (ANC) ≥ 1.5 × 10e9/L
* Platelets > 100 × 10e9/L
* Hemoglobin ≥ 9 g/dL

Hepatic Function

* AST, alanine transaminase ALT or ALP ≤ 2.5 × upper limit of normal (ULN); if liver metastases, then ≤ 5 × ULN
* Bilirubin ≤ 1.5 × ULN (< 2 × ULN if hyperbilirubinemia is due to Gilbert's syndrome)
* Serum albumin ≥ 35 g/L (3.5 g/dL)

Renal Function

* Calculated creatinine clearance of ≥ 60 mL/min by the Cockcroft-Gault equation
* Urine protein < 2+

Cardiac Function

• Left ventricular ejection fraction (LVEF) ≥ 50%

Other

* Understand and voluntarily sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)/Research Ethics Board (REB)-approved informed consent form prior to any study-specific evaluation.
* PT/PTT or INR <1.2x upper limit of normal
* Non-surgically sterile men and women of child bearing potential must agree to use highly effective methods of contraception for at least 4 months beyond the final dose received.
* Toxicity of previous antitumor therapy has returned to Grade ≤1

Exclusion Criteria:

* Patients with primary central nervous system (CNS) malignancies (Patients with stable brain metastases (≥ 4 weeks after a treatment) not requiring steroids or other treatment will be allowed on study).
* Blood transfusion within 14 days of study treatment
* Serious comorbid medical conditions such as heart, lung, kidney, liver, and brain disease that, in the opinion of the enrolling investigator, could interfere with study treatment
* Subjects with history of severe heart disease
* QTc interval using Fridericia's formula (QTcF) > 470 ms
* Estimated or known weight > 115 kg (253 lbs)
* Known/suspected pregnancy and/or lactation
* Diastolic blood pressure < 60 mmHg or >110 mmHg
* Uncontrolled intercurrent illness
* Long term care facility resident or prisoner
* Any prior receipt of a MMAE-containing drug
* Any prior receipt of a SORT1-targeting medication
* Participation in another clinical study investigating a drug or medical device or a neuro-interventional or surgical procedure that is not considered as standard care in the 30 days preceding study enrolment
* Treatment with any of the following:
* Chemotherapy or other systemic anti-cancer therapy ≤14 days or 5 half-lives (whichever is shorter) prior to first dose of study drug except for Nitrosoureas or mitomycins ≤42 days
* Major surgery ≤28 days from first dose of study drug
* Patients with a history of cerebrovascular accident within 6 months of planned first dose.
* Patients with clinically symptomatic ocular toxicities
* Patients with history of (noninfectious) interstitial lung disease (ILD)/pneumonitis that require steroids, with current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Patients with active Grade >1 peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent Adverse Events | From the time of informed consent until ~28 days after the last dose of PQ203
  The incidence and severity of Adverse Events (AEs) will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) to assess safety and tolerability.
Objective Response Rate (ORR) | From informed consent until ~28 days after the last dose of PQ203
  Tumor growth will be assessed using standard imaging techniques and scored by Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1). An Objective response rate (ORR), defined as the proportion of patients with a best overall response (BOR) of complete response (CR) or partial response (PR) will be calculated to assess preliminary signals of anti-tumor activity.

SECONDARY OUTCOMES:
Progression free survival | From informed consent to ~28 days after the last dose of PQ203
  Progression free survival (PFS; time from first dose to date of documentation of disease progression) in months will be determined.
Pharmacokinetics: Determine the Cmax of PQ203 | From first day of dosing to ~28 days after the last day of dosing
  Plasma concentration-time profiles will be used to identify the maximum drug concentration in plasma (ng PQ203/mL)
Pharmacokinetics: half-life of PQ203 in plasma | From first day of dosing until ~28 days after the last dose
  Plasma concentration-time profiles will be used to determine the half life (in hours) of PQ203 in plasma
Pharmacokinetics: PQ203 exposure | from first dose through ~28 days after the last dose
  Plasma concentration-time profiles will be used to determine the area under the curve (AUC) in ng/mL x hours
Duration of Objective Response | From Informed consent to ~28 days after the final dose
  Duration of objective response (complete or partial response) by RECIST 1.1 in months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data from PQ203-001 is planned to be shared in aggregate in a study publication.

REFERENCES:
- See also: Sponsor website — http://www.proteinqure.com/